CLINICAL TRIAL: NCT06867315
Title: Prospective, Multicenter, Randomized, Controlled, and Superiority Clinical Trial on the Safety and Effectiveness of Steep Pulse Therapy System for the Ablation of Benign Prostatic Hyperplasia
Brief Title: The Safety and Effectiveness of Steep Pulse Therapy System for the Ablation of Benign Prostatic Hyperplasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); The First Affiliated Hospital of University of Science and Technology of China (Other); First People's Hospital of Hangzhou (Other); Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Tian'an Jiang, Principal Investigator, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: steeppulse-prostate
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: steep pulse ablation
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- steep pulse therapy system (Experimental)
  Interventions: Device: steep pulse therapy system
- Tamsulosin Hydrochloride (Active Comparator)
  Interventions: Drug: Tamsulosin Hydrochloride

INTERVENTIONS:
Device: steep pulse therapy system — 1. Use steep pulse system to ablate the transitional zone of the prostate to treat BPH
  2. The steep pulse generator employs irreversible electroporation technology, which involves inserting electrodes into the tumor and delivering high-voltage electrical pulses to create nanoscale permanent pores on the lipid bilayer of tumor cell membranes. This disrupts the intracellular balance and induces cell apoptosis
  Arms: steep pulse therapy system
Drug: Tamsulosin Hydrochloride — 1. use Tamsulosin Hydrochloride Sustained-Release Capsules to treat BPH
  2. the brand name is Harnal®
  3. the specification is 0.2mg per capsule
  Arms: Tamsulosin Hydrochloride

SUMMARY:
The goal of this clinical trial is to assess the efficacy of steep pulse ablation in treating benign prostatic hyperplasia (BPH) and to evaluate its safety profile in treating BPH. The main questions it aims to answer are:

1. whether steep pulse ablation can effectively manage BPH symptoms and to investigate any potential safety concerns associated with its use in treating BPH.
2. If steep pulse ablation can perform superior effect than Tamsulosin Hydrochloride in treating BPH.

Participants will be asked to do:

1. Participants will be given Tamsulosin Hydrochloride or undergo steep pulse ablation.
2. Participants will be followed up after 1 month and 3 month after taking drug or undergo ablation for test and relative examinations.

ELIGIBILITY:
Inclusion Criteria:

1. patients with BPH diagnosed through digital rectal examination, B-mode ultrasound and urinary flow rate.
2. international prostate symptom score(IPSS)>=12.
3. Maximum urinary flow rate between >5ml/s and <15ml/s with a minimum voided volume ≥ 150ml.
4. Age ≥ 50 years old.
5. Subjects are willing to participate and have signed the informed consent form.

Exclusion Criteria:

1. Patients with acute or severe urinary tract infections.
2. Patients clinically diagnosed with prostate cancer.
3. Patients with neurogenic bladder or bladder dysfunction due to other factors.
4. Patients with urethral stricture.
5. Patients who have undergone previous prostatectomy (TURP), enucleation, or laser surgery.
6. Patients with implanted pacemakers or metal replacements in the pelvis or hip joints.
7. Patients who cannot tolerate general anesthesia or surgery due to severe systemic diseases, heart diseases, pulmonary insufficiency, failure of vital organs, or other reasons.
8. Patients in the trial group who have taken medications that can affect BPH symptoms within 3 months of postoperative follow-up.
9. Patients who have participated in other drug trials or medical device clinical trials within 3 months prior to enrollment.
10. Patients deemed unsuitable for participation in this clinical trial by the investigator.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
The change in maximum urinary flow rate | 3 months
  compare the maximum urinary flow rate of the patients post treatment to the baseline level of the patients

SECONDARY OUTCOMES:
changes in the international prostate symptoms score(IPSS) before and after treatment | screening, 30 days and 3 months
  compare the IPSS of the patients in screening stage, 30 days after treatment and 3 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China